CLINICAL TRIAL: NCT02511197
Title: Safety and Diagnostic Performance of 68Ga-NOTA-PRGD2 PET/CT in Patients With Lung Injury and Pulmonary Fibrosis
Brief Title: 68Ga-NOTA-PRGD2 PET/CT in Patients With Lung Injury and Pulmonary Fibrosis
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PUMCHNM10
Record Dates: First submitted 2015-07-23; First posted 2015-07-29 (Estimated); Last update posted 2017-04-06 (Actual); Status verified 2015-07

CONDITIONS: Pulmonary Fibrosis, Unspecified
Keywords: PET; lung injury; integrin receptor
MeSH Terms: conditions — Pulmonary Fibrosis; Lung Injury | interventions — Positron Emission Tomography Computed Tomography

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 68Ga-NOTA-PRGD2 injection & PET/CT scan (Experimental): The patients were intravenously injected with 68Ga-NOTA-PRGD2 in one dose in nearly 111 MBq and then underwent PET/CT scan 0.5 h later.
  Interventions: Drug: 68Ga-NOTA-PRGD2; Device: PET/CT

INTERVENTIONS:
Drug: 68Ga-NOTA-PRGD2 — 68Ga-NOTA-PRGD2 were injected into the patients before the PET/CT scans
  Other Names: 68Ga-NOTA conjugated with dimer PRGD2
Device: PET/CT

SUMMARY:
This is an open-label positron emission tomography/computed tomography (PET/CT) study to investigate the diagnostic performance and evaluation efficacy of 68Ga-NOTA-PRGD2 in lung injury (LI) and pulmonary fibrosis (PF) patients. A single dose of nearly 111 MBq 68Ga-NOTA-PRGD2 (≤ 40 µg NOTA-PRGD2) will be intravenously injected into patients with LI/PF. Visual and semiquantitative method will be used to assess the PET/CT images.

DETAILED DESCRIPTION:
The αvβ3-integrin is a transmembrane heterodimeric receptor that mediates cell-cell and cell-extracellular matrix adhesion. The αvβ3-integrin plays a pivotal role in promoting and sustaining angiogenesis and fibrosis. Cyclic arginine-glycine-aspartic acid (RGD) peptide is the key integrin recognition motif that can strongly bind to the αvβ3-integrin, which makes the RGD-based peptides hold a promise for imaging and treatment of diseases characterised with angiogenesis and fibrosis including LI and PF.

Animal study in bleomycin induced lung fibrosis showed good uptake ratio of 68Ga-NOTA-PRGD2 in lung vs background. For interests in clinical translation of 68Ga-NOTA-PRGD2, an open-label dynamic whole-body PET/CT study was designed to investigate safety and diagnostic performance of 68Ga-NOTA-PRGD2 in patients with LI or PF.

ELIGIBILITY:
Inclusion Criteria:

Patients with idiopathic pulmonary fibrosis

* Males and females, ≥18 years old.
* Characteristic clinical signs, symptoms and laboratory tests suggesting the diagnosis of LI/PF.
* The diagnosis of IPF is based on The Centres for Disease Control and Prevention (CDC) criteria for diagnosing LI/PF. They rely on a combination of clinical, radiological, operative and histological findings, in addition to results of other laboratory tests.

Exclusion Criteria:

* Females planning to bear a child recently or with childbearing potential.
* Renal function: serum creatinine >3.0 mg/dL (270 μM/L).
* Liver function: any hepatic enzyme level more than 5 times upper limit of normal.
* Known severe allergy or hypersensitivity to IV radiographic contrast.
* Patients not able to enter the bore of the PET/CT scanner.
* Inability to lie still for the entire imaging time because of cough, pain, etc.
* Inability to complete the needed examinations due to severe claustrophobia, radiation phobia, etc.
* Concurrent severe and/or uncontrolled and/or unstable other medical disease that, in the opinion of the investigator, may significantly interfere with study compliance.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2015-05; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Visual assessment of lung lesions | 1 year
  Visual analysis will be performed by consensus reading by at least 3 experienced nuclear medicine physician.
Semiquantitative assessment of lung lesions | 1 year
  The semiquantitative analysis will be performed by the same person for all the cases, and the standardized uptake values (SUVs) of lungs will be measured.

SECONDARY OUTCOMES:
Adverse events collection | 5 days
  Adverse events within 5 days after the injection and scanning of patients and patients will be followed and assessed.
Routine blood test | 24 hours
  Routine blood test of healthy volunteers will be measured before injection and 24 hours after test.
Serum albumin | 24 hours
  Serum albumin of healthy volunteers will be measured before injection and 24 hours after test.
Routine urine test | 24 hours
  Routine urine test of healthy volunteers will be measured before injection and 24 hours after test.

CONTACTS AND LOCATIONS:
Overall Officials: Zhaohui Zhu, MD, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, China